CLINICAL TRIAL: NCT02845323
Title: Randomized Phase II Study of Neoadjuvant Nivolumab With and Without Urelumab in Cisplatin-Ineligible or Chemotherapy-refusing Patients With Muscle-Invasive Urothelial Carcinoma of the Bladder
Brief Title: Neoadjuvant Nivolumab With and Without Urelumab in Cisplatin-Ineligible or Chemotherapy-refusing Patients With Muscle-Invasive Urothelial Carcinoma of the Bladder
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J1682; IRB00103062 (Other: JHMIRB)
Record Dates: First submitted 2016-07-13; First posted 2016-07-27 (Estimated); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Urothelial Carcinoma; Bladder Cancer
MeSH Terms: conditions — Carcinoma, Transitional Cell; Urinary Bladder Neoplasms | interventions — Nivolumab; urelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nivolumab in combination with Urelumab (Experimental): Nivolumab and Urelumab combination:
  Nivolumab 240 mg will be administered by 1 hour intravenous infusion on day 1 and day 15 for two cycles
  Urelumab 8mg will be administered by 1 hour intravenous infusion on day 1 for two cycles
  Interventions: Drug: Nivolumab in combination with Urelumab
- Nivolumab monotherapy (Active Comparator): Nivolumab 240 mg will be administered by 1 hour intravenous infusion on day 1 and day 15 for two cycles
  Interventions: Drug: Nivolumab monotherapy

INTERVENTIONS:
Drug: Nivolumab in combination with Urelumab — Two cycles of Nivolumab Two cycles of Urelumab
  Other Names: Opdivo
  Arms: Nivolumab in combination with Urelumab
Drug: Nivolumab monotherapy — Two cycles of Nivolumab alone
  Arms: Nivolumab monotherapy

SUMMARY:
This study evaluates the post cystectomy CD8+ tumor response of patients receiving Nivolumab plus Urelumab versus Nivolumab alone. Half the patients will receive Nivolumab plus Urelumab, while the other half will receive Nivolumab alone.

DETAILED DESCRIPTION:
This is phase II clinical trial design randomizing patients who are cisplatin-ineligible or chemotherapy-refusing with MIBC (stages T2-T4, N0-N2, M0) to one of two treatment arms: Arm A - Nivolumab in combination with Urelumab or Arm B - Nivolumab monotherapy.

The study population will include male and female patients over the age of 18 with muscle invasive urothelial carcinoma of the bladder (MIBC) who are not suitable for cisplatin-based chemotherapy or refuse chemotherapy, but are fit to undergo surgical resection of their cancer by cystectomy. Patients with resectable clinical node positive disease within the true pelvis are eligible.

ELIGIBILITY:
Inclusion Criteria:

* Electively refusing cisplatin-based neoadjuvant chemotherapy or
* Ineligible to receive cisplatin-based neoadjuvant chemotherapy based upon at least one of the following criteria:
* Creatinine clearance < 60 ml/min
* ECOG status =2
* Grade > 2 hearing loss
* Grade > 2 neuropathy
* New York Heart Association Class III heart failure
* Age ≥ 18 years old at time of consent
* Patients must have the following laboratory values:

  a) Absolute neutrophil count (ANC) ≥ 1.5 K/mm3 (must be stable off any growth factor within 4 weeks of first study drug administration) b) Platelets ≥ 100 K/mm3 (transfusion to achieve this level is not permitted within 2 weeks of first study drug administration) c) Hemoglobin (Hgb) ≥ 9 g/dL d) Serum total bilirubin: ≤ 1.5 x ULN e) ALT and AST ≤ 3.0 x ULN f) Serum creatinine clearance (CrCl) ≥ 30 mL/min using the Cockcroft-Gault equation, see formula below:
* CrCl = [140-age (years)] x weight (kg) / [72 x serum Cr (mg/dL)] (if patient is female multiply the above by 0.85)
* Patients who give a written informed consent obtained according to local guidelines

Exclusion Criteria:

* Patients with locally advanced unresectable or metastatic urothelial carcinoma as assessed on baseline radiographic imaging obtained within 28 days prior to study registration. The required radiographic imaging includes:

  a) Abdomen/Pelvis - CT scan b) Chest - chest x-ray or CT scan
* Patients with concurrent upper urinary tract (i.e. ureter, renal pelvis) invasive urothelial carcinoma.
* Patients with another active second malignancy other than non-melanoma skin cancers and biochemical relapsed prostate cancer
* Patients who have received the last administration of an anti-cancer therapy including chemotherapy, immunotherapy, and monoclonal antibodies ≤ 4 weeks prior to starting study drug, or who have not recovered from the side effects of such therapy
* Patients who have received prior therapy with immune checkpoint inhibitors (e.g. anti-PD-1, anti-PD-L1, anti-LAG3, anti-CTLA-4) or immune costimulatory molecules (e.g. anti-CD137, anti-OX40, anti-GITR) directed agents.
* Patients who have had radiotherapy ≤ 4 weeks prior to starting study drug, or who have not recovered from radiotherapy toxicities
* Patients who have undergone major surgery (e.g. intra-thoracic, intra-abdominal or intra-pelvic), open biopsy or significant traumatic injury ≤ 4 weeks prior to starting study drug, or patients who have had minor procedures (i.e. TURBT), percutaneous biopsies or placement of vascular access device ≤ 1 week prior to starting study drug, or who have not recovered from side effects of such procedure or injury
* Patients with history of alcoholic or non-alcoholic steatohepatitis (NASH), auto-immune hepatitis, or previous grade 3-4 drug-related hepatitis. (Note: Patients with radiographic evidence of steatohepatitis are excluded unless a liver biopsy is obtained demonstrating no evidence of alcoholic or non-alcoholic steatohepatitis).
* Patient with history of prior solid organ or allogeneic bone marrow transplant.
* Patients with any of the following concurrent severe and/or uncontrolled medical conditions which could compromise participation in the study:

  1. Clinically significant cardiac diseases, including any of the following:

  i. History or presence of serious uncontrolled ventricular arrhythmias

ii.Clinically significant resting bradycardia

iii.Any of the following within 3 months prior to starting study drug: myocardial infarction (MI), severe/unstable angina, Coronary Artery Bypass Graft (CABG), Congestive Heart Failure (CHF), Cerebrovascular Accident (CVA), Transient Ischemic Attack (TIA), Pulmonary Embolism (PE)

iv.Uncontrolled hypertension defined by a SBP ≥ 160 mm Hg and/or DBP ≥ 100 mm Hg, with or without anti-hypertensive medication(s)

b) Cirrhosis, chronic active hepatitis or chronic persistent hepatitis

c) Known diagnosis of human immunodeficiency virus (HIV) infection (HIV testing is not mandatory)

d) Known diagnosis of any condition (i.e. post-hematopoietic or organ transplant, rheumatoid arthritis, systemic lupus erythematosus, inflammatory bowel disease, etc.) that requires chronic immunosuppressive therapy. Usage of non-steroidal anti-inflammatory medications (NSAIDS) for the treatment of osteoarthritis and uric acid synthesis inhibitors for the treatment of gout are permitted. For questions, please consult the study chair.

e) Other concurrent severe and/or uncontrolled concomitant medical conditions (e.g. active or uncontrolled infection, uncontrolled diabetes) that could cause unacceptable safety risks or compromise compliance with the protocol

* Pregnant or breast-feeding women
* Women of child-bearing potential, who are biologically able to conceive, and not employing two forms of highly effective contraception. Highly effective contraception must be used throughout the trial and up to 8 weeks after the last dose of study drug (e.g. male condom with spermicidal; diaphragm with spermicide; intra-uterine device). Women of child-bearing potential, defined as sexually mature women who have not undergone a hysterectomy or who have not been naturally postmenopausal for at least 12 consecutive months (i.e., who has had menses any time in the preceding 12 consecutive months), must have a negative serum pregnancy test ≤ 14 days prior to starting study drug
* Fertile males not willing to use contraception, as stated above
* Patients unwilling or unable to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-05-16 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Immune response to treatment with Nivolumab and Urelumab compared to Nivolumab monotherapy measured by tumor infiltrating CD8+ T cell density at cystectomy | 2 years

SECONDARY OUTCOMES:
To evaluate the number of participants with treatment-related adverse events as assessed by CTCAE v 4.0 | 2 years
Proportion of patients achieving pathologic response (<pT2N0) with Nivolumab and Urelumab and the use of Urelumab alone | 2 years
Prognostic value of tumor biopsy PD-1 and PD-L1 expression and change in expression for pathologic tumor response as defined by cystectomy pathologic staging <pT2 N0 in patients treated with Nivolumab | 2 years
Change in expression for pathologic tumor response as defined by cystectomy pathologic staging <pT2 N0 in patients treated with Nivolumab | 2 years
Prognostic value of tumor bx 4-1BB (CD137)& 4-1BB ligand (CD137L) expression | 2 years
Change in expression, assessed by (IHC) analysis, for tumor response, defined by cystectomy staging < pT2N0, in cisplatin-ineligible MIBC pts tx w/Urelumab. | 2 years
Prognostic value of tumor biopsy 4-1BB expression | 2 years
Change in expression, assessed by (IHC) analysis, for pathologic CR response, defined by cystectomy staging pT0N0, in cisplatin-ineligible MIBC pts tx w/ Urelumab. | 2 years
Proportion of patients achieving pathologic complete response with neoadjuvant Nivolumab and Urelumab (Arm A) and Nivolumab monotherapy (Arm B). | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Noah Hahn, MD, Principal Investigator — Johns Hopkins University
Locations (5):
- United States (5):
  - UCLA Institute of Urologic Oncology, Los Angeles, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - University of Chicago, Chicago, Illinois
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Columbia University Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: No